CLINICAL TRIAL: NCT03596684
Title: Citrulline Efficacy to Improve Carbohydrate Metabolism Abnormalities in the Patient Treated With High Doses of Statin
Acronym: STATIMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 69HCL17_0754; 2018-A00575-50 (Other: ID-RCB)
Record Dates: First submitted 2018-06-04; First posted 2018-07-24 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Atorvastatin
Keywords: Carbohydrate Metabolism; Citrulline; Statine
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- citrulline (Experimental): citrulline 5g/d
  Interventions: Dietary Supplement: citrulline supplementation; Procedure: glucose tolerance test
- Placebo (Placebo Comparator): pure mixture of amino acids: alanine, aspartate, glycine, proline, serine, histidine
  Interventions: Dietary Supplement: placebo supplementation; Procedure: glucose tolerance test

INTERVENTIONS:
Dietary Supplement: citrulline supplementation — 2.5 g per os of citrulline on the morning and the evening (5 g/ jour) during 4 weeks.
  Arms: citrulline
Dietary Supplement: placebo supplementation — 2.5 g of the product in the morning and in the evening during 4 weeks.
  Arms: Placebo
Procedure: glucose tolerance test — 2 exploration mornings distant from 28 days (before and after citrulline) will allow carrying out an oral glucose tolerance test of 2 hours (75 g glucose per os)

SUMMARY:
Hypercholesterolemia is a major cardiovascular risk factor. Statins are the first-line drug treatment for hypercholesterolemia and have been shown to be effective in both primary and secondary prevention of cardiovascular disease. However, long-term statin therapy is associated with impaired carbohydrate metabolism and increased risk of developing type 2 diabetes (T2D), particularly in patients with metabolic syndrome. The risk of developing T2D is higher with high doses of statins.

Currently the benefits of statins on the reduction of major cardiovascular events and mortality are considered superior to the risk of statin-induced diabetes T2D, and no change in clinical practice has been recommended to date. However, it now appears necessary to develop strategies to reduce the adverse effects of statins on carbohydrate metabolism and maintain the carbohydrate tolerance of patients on statins, especially in those at risk of developing T2D under statins.

Statins are able to induce the expression and activity of an enzyme synthesizing nitric oxide (NO), the endothelial NO synthase (eNOS), which helps improving insulin sensitivity and insulin secretion. However, availability and metabolism of its substrate arginine is impaired in obesity and T2D. The investigators thus hypothesized that providing citrulline to statin treated patients, the arginine precursor with better gastrointestinal tolerance and bioavailability than arginine, would beneficially impact their glucose homeostasis.

Tested in vivo by Béatrice Morio, a member of the CarMeN laboratory, combining citrulline to atorvastatin improved glucose tolerance and insulin sensitivity in mice fed a high fat-high sucrose diet. These data therefore suggest that combining citrulline to atorvastatin may improve glucose tolerance in statin-treated patients at high risk of developing T2D.

The objective of the study is therefore to investigate the impact of citrulline supplementation (5g/d) vs. placebo for 4 weeks on glucose tolerance assessed during an oral glucose tolerance test in patients at risk for developing T2D and treated with atorvastatin (40 or 80 mg / day).

ELIGIBILITY:
Inclusion Criteria:

* 40 years old < Age <75 years old
* men and women who are menopausal or who benefit from effective contraception
* treatment with atorvastatin at 40 or 80 mg / d for more than 3 months for primary prevention or secondary prevention at more than 3 months of the acute event (stroke, acute coronary syndrome) with or without ezetimibe (Ezetrol® monotherapy or in the form of associated with atorvastatin Liptruzet® 10/40 or 10/80)
* with a Body Mass Index (BMI) ≥28 kg / m2 and at least one other risk factor for statin-dependent diabetes among the following 4:

  * Blood pressure ≥ 140/90 mmHg or hypotensive treatment
  * Triglyceridemia ≥ 150 mg / l
  * Fasting blood glucose ≥ 100 mg / dl
  * HDL-cholesterol <40 mg / dL in men, <50 mg / dL in women
* affiliated to a social security scheme
* signed informed consent

Exclusion Criteria:

- General criteria:

* Subject with unstable medical or psychological conditions that, in the opinion of the investigator, could lead the subject to be non-compliant or uncooperative during the study or could compromise the safety or participation of the subject under study L.1121-6, L.1121-8, L.1121-9 and L1122-1-2 of the Public Health Code).
* Major subjects under guardianship or deprived of their liberty by judicial or administrative decision.
* Plan for weight loss during the previous 3 months, current or future
* Dietary supplements for weight loss (based on plant extracts, algae, pre- and probiotics) in the previous 3 months or in progress

Biological criteria:

* Aspartate Amino Transferase (ASAT), Alanine Amino Transferase (ALAT)> 2 times the normal values
* HbA1c> 6.5%
* Creatin Phospho Kinase (CPK)> 2 times normal
* Triglycerid > 5g / L
* Renal insufficiency (clearance <60 mL / min)
* Demonstration of a biological abnormality deemed by the investigator to be clinically significant

Medical and therapeutic criteria:

* Diabetes type 1 or 2
* Subjects treated with a drug that may interfere with the metabolism of citrulline and glucose (vitamin K antagonists, corticosteroids for more than 8 days before the study, anorexigenic drugs (Anorex, Fenproporex Deglaude AP, Moderatan, Prefamone Chronules), drugs (Orlistat, Lioresal)
* Any associated or uncontrolled progressive pathology (cardiac pathology, myocardial infarction of less than 6 months, arterial hypertension, psychiatric, renal or hepatic, cancer).
* pregnant or lactating woman
* Consumption of more than 3 glasses of alcohol per day.
* Subjects who express any reluctance to consume a food supplement morning and evening.
* eating disorders.
* Weight variation of +/- 5% during the previous 3 months
* Severe, progressive affection.
* Depressive or psychiatric state (antidepressant or psychotropic treatment).
* Medical or surgical history deemed by the investigator to be incompatible with this study.
* Blood donation in the 2 months prior to inclusion.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
difference in the area under the curve of the glycemic response during a 75 g glucose tolerance test between the end and the beginning of citrulline supplementation versus placebo | 4 weeks

SECONDARY OUTCOMES:
Difference in the index of insulin sensitivity determined during Oral Glucose Tolerance Test (OGTT) performed at the end and before the supplementation in citrulline versus placebo | 4 weeks
Difference in the index of insulin secretion determined during OGTT performed at the end and before the supplementation in citrulline versus placebo | 4 weeks
occurrence of adverse events and serious adverse events for assessment of tolerability | assessed up 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Charriere, MD, Principal Investigator — Hospices Civils de Lyon Endocrinology and diabetology service, Louis Pradel Hospital
Locations (1):
- Endocrinology and diabetology service, Louis Pradel Hospital, Bron, France